CLINICAL TRIAL: NCT02843958
Title: Validation of a Portable Medical Device for Diagnostic in Vitro, Designed to Measure Blood Coagulation's Biological Parameters
Brief Title: Validation of a Portable Medical Device for Diagnostic in Vitro
Acronym: HEMOPTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 38RC14.008
Record Dates: First submitted 2016-07-12; First posted 2016-07-26 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Volunteer; Patients Under Vitamin K Antagonist (VKA)
Keywords: Medical device; Hemoptic; Vitamin K antagonist; Diagnostic in vitro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers and patients under Vitamin K antagonist (Other)
  Interventions: Device: HEMOPTIC

INTERVENTIONS:
Device: HEMOPTIC

SUMMARY:
This clinical trial is about a new technology, named HEMOPTIC. It enables to mesure time of blood coagulation for monitoring of patients under Vitamin K antagonist (VKA).

This device was created as an alternative to blood sample, that have to be done in a medical laboratory.

The main goal is to evaluate the accuracy of the International Normalized Ratio (INR) measurement of this new portable device for diagnostic in vitro, among healthy patients and patients under anti-vitamin K treatment.

ELIGIBILITY:
Inclusion Criteria of healthy volunteers:

* Man or woman between 18 and 70 years
* Body Mass Index >18 and <29
* Absence of any acute pathology in the month preceding the study
* To be affiliated or beneficiary of social security

Exclusion Criteria of healthy volunteers:

* Pregnant, partutient or breastfeeding woman
* Patient with Raynaud's syndrome
* Person deprived of liberty by legal or administrative decision, person to a legal protection order
* Deferral periods for other clinical studies
* Annual threshold compensation attain for biomedical search participations

Inclusion Criteria of patients:

* Man or woman between 18 and 80 years
* Patient treated by oral anti vitamin K anticoagulants (coumadine, warfarine, fluidione)
* Absence of any acute pathology in the month preceding the study
* To be affiliated or beneficiary of social security

Exclusion Criteria of healthy patients:

* Pregnant, partutient or breastfeeding woman
* Patient with Raynaud's syndrome
* Person deprived of liberty by legal or administrative decision, person to a legal protection order
* Deferral periods for other clinical studies
* Annual threshold compensation attain for biomedical search participations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
International Normalized Ratio measurement: comparison to the standard reference. | V2

SECONDARY OUTCOMES:
International Normalized Ratio measurement: repeatability | V2
International Normalized Ratio measurement:reproductibility | V2

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Cracowski, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Heneghan C, Alonso-Coello P, Garcia-Alamino JM, Perera R, Meats E, Glasziou P. Self-monitoring of oral anticoagulation: a systematic review and meta-analysis. Lancet. 2006 Feb 4;367(9508):404-11. doi: 10.1016/S0140-6736(06)68139-7. PMID 16458764
- [Background] Faivre M, Peltie P, Planat-Chretien A, Cosnier ML, Cubizolles M, Nougier C, Negrier C, Pouteau P. Coagulation dynamics of a blood sample by multiple scattering analysis. J Biomed Opt. 2011 May;16(5):057001. doi: 10.1117/1.3573813. PMID 21639579
- [Background] Matchar DB, Jacobson A, Dolor R, Edson R, Uyeda L, Phibbs CS, Vertrees JE, Shih MC, Holodniy M, Lavori P; THINRS Executive Committee and Site Investigators. Effect of home testing of international normalized ratio on clinical events. N Engl J Med. 2010 Oct 21;363(17):1608-20. doi: 10.1056/NEJMoa1002617. PMID 20961244
- [Background] McBride GB (2005) A proposal for strength-of-agreement criteria for Lin's Concordance Correlation Coefficient. NIWA Client Report: HAM2005-062.
- [Background] Riberolles, C. (2009). Résultats du PHRC autocontôle de l'anticoagulation. Conférence. XIXes Journées européennes de la Société française de cardiologie, Paris.